CLINICAL TRIAL: NCT02663492
Title: Transcutaneous Electrical Acupoint Stimulation Ameliorates Chemotherapy-Induced Bone Marrow Suppression in Lung Cancer Patients
Brief Title: Transcutaneous Electrical Acupoint Stimulation for Non-small Cell Lung Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji University (Other)
Responsible Party: Principal Investigator, Caicun Zhou, Director, Tongji University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TEAS_001
Record Dates: First submitted 2016-01-15; First posted 2016-01-26 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Non-Small Cell Lung Cancer; Lung Cancer
Keywords: Acupuncture; electrical stimulation of acupoints; chemotherapy; Diyu Shengbai Pian; nursing care
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TEAS group (Experimental): Patients with transcutaneous electrical acupoint stimulation (TEAS) group receive electrical stimulation of acupoints including Dazhui (DU14), Geshu (BL17), Zusanli (ST36), Sanyinjiao (SP6), and Hegu (LI4).
  Interventions: Device: TEAS
- Medication group (Active Comparator): On the basis of routine nursing care, patients need to take Sanguisorba officinalis L., named Diyu Shengbai Pian (a Traditional Chinese Medicine) 3 times per day.
  Interventions: Drug: Sanguisorba officinalis L.
- Control group (No Intervention): The patients of control group receive routine nursing care, including (1) to be observed the changes in patient condition, (2) to eat high-calories, high-protein, high-vitamin, easy-to-digest foods during chemotherapy, (3) to be treated by psychological care, (4) to be prevented against the occurrence of phlebiti, and (5) to use Ondansetron and Omeprazole as direction.

INTERVENTIONS:
Device: TEAS — The patients will be treated by their assigned acupuncture stimulation in 7 days. The surface electrical stimulation devices and application parameter are: G6805-II pulse acupuncture treatment instrument from Shanghai Medical Technology Company, Ltd (Shanghai, China); sparse-dense wave stimulation (sparse wave 30Hz; dense wave 100Hz) with an intensity of 6-15 V; and the corresponding parts of the body experienced a slight quiver, with a duration 20 minutes each time.
  Arms: TEAS group
Drug: Sanguisorba officinalis L. — Sanguisorba officinalis L., a Leukogenic medication, named Diyu Shengbai Pian (Chengdu Diao Tianfu Pharmaceutical Group Co., Ltd., China) will be taken 0.4g each time by 3 times per day.
  Other Names: Diyu Shengbai Pian
  Arms: Medication group

SUMMARY:
To investigate the effect of percutaneous electrical stimulation on chemotherapy-induced bone marrow suppression in patients with lung cancer.

DETAILED DESCRIPTION:
Lung cancer is the malignant neoplasm with the highest incidence and mortality in China as well as worldwide. Non-small cell lung cancer (NSCLC) accounts for 80%-85% of all lung cancer cases. Chemotherapy is the preferred treatment method for NSCLC, but many patients cannot tolerate the adverse reactions of chemotherapy. Among the most common and most severe adverse reactions is bone marrow suppression. The more serious the bone marrow suppression, the higher the direct medical cost of chemotherapy. Literatures showed Acupuncture was used to treat patients with chemotherapy-induced bone marrow suppression. In this study, the effect of percutaneous electrical stimulation of acupoints including Dazhui (DU14), Geshu (BL17), Zusanli (ST36), Sanyinjiao (SP6), and Hegu (LI4) will be investigated, compared with the medication group treated by oral administration of prophylactic agents, and the control group received routine nursing care on chemotherapy-induced bone marrow suppression in patients with lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Non-small cell lung cancer(NSCLC)
* age between 20 and 75 years
* chemotherapy naive after diagnosis
* GP regimen as treatment
* an expected survival of more than 12 weeks based on a score equal to or greater than 60 points on Karnofsky performance status (KPS) scale
* the ability to understand and speak Mandarin

Exclusion Criteria:

* diagnosis of a hematological system tumor
* mental illness
* bone marrow suppression prior to chemotherapy
* pregnancy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-01 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change of Blood routine indexes in 1 month | Day 0, Day 5, Day 8, Day 11, Day 14, Day 21 and Day 28
  The routine blood examinations of indicators of bone marrow suppression, including red blood cells (10^12/L), hemoglobin (g/L), white blood cells (10^9/L), and platelets (10^9/L).

SECONDARY OUTCOMES:
Change of Comfort Degree | Day 0, Day 8, and Day 28
  The Comfort Scale is assessed using General Comfort Questionnaire designed by KY Kolcaba. A preliminary experiment was conducted in 30 patients with NSCLC before the first visit, and the reliability coefficient of the scale was calculated; Cronbach's alpha = 0.932 indicated high internal consistency.

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, Doctor, Principal Investigator — Shanghai Pulmonary Hospital of Tongji University, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital Medical Oncology Department, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No